CLINICAL TRIAL: NCT01147328
Title: Assessing the Impact of Health Information Exchange (HIE) on Healthcare Utilization
Acronym: VHR
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0708160258-08
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Health Information Technology; Health Information Exchange; Virtual Health Record; Health Care Utilization
Keywords: Health information technology; Health information exchange; Virtual health record; Health care utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients who did not have their data accessed in the VHR by a provider within 6 months after they consented will be part of the control group
  Interventions: Other: Virtual Health Record (VHR)
- 2: Patients who had their data accessed in the VHR by a provider within 6 months after they consented will be part of the intervention group
  Interventions: Other: Virtual Health Record (VHR)

INTERVENTIONS:
Other: Virtual Health Record (VHR) — Technology that enables providers to electronically access community-wide clinical data for patients who have consented to have their clinical data accessed via a web portal.

SUMMARY:
The purpose of this study is to assess usage of the virtual health record (VHR), and determine the effects of this technology on healthcare utilization.

DETAILED DESCRIPTION:
National efforts are underway to support the implementation of technology that enables providers to electronically access and view community-wide clinical information for their patients, which has the potential to improve quality of care and reduce health care costs by providing timely and complete health information at the point of care. However, few empirical studies have been conducted to evaluate the economic effects of this technology. Along with other stakeholders, New York State is funding regional health information organizations (RHIOs) to deploy a virtual health record (VHR), which is technology that enables providers to electronically access community-wide clinical data for patients who have consented to have their clinical data accessed via a web portal. RHIOs bring together multiple stakeholders, including physician practices, hospitals, pharmacies, and laboratories, for the purpose of exchanging clinical information electronically across communities. The investigators will conduct a multi-RHIO retrospective pre-post, cohort study of adult patients who have consented to have their clinical data viewed by their providers using the VHR portal. Examining the effects of electronically accessing clinical data on healthcare utilization across multiple settings and communities can help inform the national health IT initiative that is underway and allow assessment of the economic value of these technologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are aged 18 and older who have consented during the year 2009 to allow their provider use of their VHR data and had at least one visit to a healthcare provider that is a VHR user within 6 months after they consented to allow their provider use of their VHR data. (Note: we only wish to include individuals who have had the opportunity for their data to be viewed using the VHR web portal). Providers who are participating in the Regional Health Information Exchange (RHIO).

Exclusion Criteria:

* Patients and providers who do not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with concurrent controls who have consented to have their clinical data viewed by their providers using the VHR portal provided by RHIOs. Providers who are participating in the Regional Health Information Exchange (RHIO).
Sampling Method: Non-Probability Sample
Enrollment: 218766 (Actual)
Dates: Start 2011-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
VHR Usage | 1 year
  Data from the VHR web portal database which records patient consent and provider usage of the web portal
Changes in Healthcare Utilization | 1 year
  A retrospective set of claims data will be used to characterize healthcare utilization and describe the study population

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Kern, MD, MPH, Study Chair — Weill Medical College of Cornell University; Yolanda Barron, MS, Study Chair — Weill Medical College of Cornell University; Alison Edwards, MStat, Study Chair — Weill Medical College of Cornell University; Ranjit Singh, MD, MA, MBA, Study Chair — Weill Medical College of Cornell University; Renny Varghese, MPH, Study Chair — Weill Medical College of Cornell University; Vaishali Patel, PhD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - HealtheLink, Buffalo, New York
  - Weill Medical College of Cornell University, New York, New York
  - Rochester RHIO, Rochester, New York